CLINICAL TRIAL: NCT05818280
Title: Relationship Between 24-hour Blood Pressure Variability and FRagility in the Elderly Patient
Acronym: VAR-24hFR
Status: Completed | Type: Observational
Sponsor: Pr. Nicolas GIRERD (Other)
Responsible Party: Sponsor-Investigator, Pr. Nicolas GIRERD, Study chair, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2022PI197
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: Hypertension; Frail patient
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In the 2016's Haute Autorité de Santé (HAS) recommendations (Haute Autorité de Santé. Management of arterial hypertension in adults. Saint-Denis La Plaine: HAS; 2016.) concerning the management of arterial hypertension in adults, the Ambulatory Blood Pressure Measurement (ABPM) is described as a diagnostic tool for hypertension as well as a tool useful for checking blood pressure (BP) control in treated patients.

It is also stipulated that ABPM can provide additional information such as the exploration of significant blood pressure variability.

The 2014's ESH recommendations (ESH practical guidelines for ambulatory blood pressure monitoring, 2014) concerning ABPM indicate that variability of BP over 24 hours can be considered as a research parameter.

Blood Pressure Variability could be a better predictor of organ damage related to hypertension than blood pressure measured in consultation.

Furthermore, BP measurement over 24 hours has been demonstrated as a more sensitive risk factor for cardiovascular events such as stroke or ischemic coronary events.

It is specified in the 2018 ESH/ESC guidelines on the management of hypertension (Mancia G, et al. 2018 ESC/ESH Guidelines for the management of arterial hypertension. 2018) that an additional number of ABPM parameters may have prognostic value such as 24-hour variability even if there is no indication yet of its evaluation in clinical routine.

The variability of blood pressure is associated with an increased risk of cardiovascular events, in particular stroke and coronary events in young and hypertensive patients, regardless of their cardiovascular risk factors, mean value of their systolic BP measured in ABPM or during consultation follow-up as shown by Rothwell PM et al. (Prognostic significance of visit-to-visit variability, maximum systolic blood pressure, and episodic hypertension. The Lancet. mars 2010;375(9718):895-905) and Mehlum MH et al. (Blood pressure variability and risk of cardiovascular events and death in patients with hypertension and different baseline risks. Eur Heart J. 21 juin 2018;39(24):2243-51.)

Studies also show that BP variability in elderly hypertensive patients is an independent risk factor for cardiovascular events (Eto M et al. Impact of Blood Pressure Variability on Cardiovascular Events in Elderly Patients with Hypertension. Hypertens Res. 2005;28(1):1-7.) and that BP variability would be greater in the elderly patient (Magdás A et al. Ambulatory monitoring derived blood pressure variability and cardiovascular risk factors in elderly hypertensive patients. Biomed Mater Eng. 2014;24(6):2563-9)

Finally, a link between frailty and blood pressure variability is demonstrated by Rouch L et al. (Visit-to-Visit Blood Pressure Variability and Incident Frailty in Older Adults. Le Couteur D, éditeur. J Gerontol Ser A. 13 juill 2021;76(8):1369-75.) However, BP variability, measured in this study by blood pressure variation between clinical visits, does not assess overnight variability. Another limitation in the evaluation of frailty is the exclusion of patients with an MMSE < 24.

Hussain SM et al. (Variation in Mean Arterial Pressure Increases Falls Risk in Elderly Physically Frail and Prefrail Individuals Treated With Antihypertensive Medication. Hypertension. sept 2022;79(9):2051-61.) also show that BP variability measured by ABPM would increase the risk of serious falls in frail or pre-frail elderly subjects taking antihypertensive treatment.

The objective of this study is therefore to evaluate the link between blood pressure variability on 24-hour recordings measured by the standard deviation and the coefficient of variation, according to the frailty status in patients aged over 75 with hypertension, treated or not with antihypertensive molecules.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 75 years old, men and women,
* Patients admitted for consultation or day hospitalisation to the Geriatric Service of the CHRU, living at home, with treated or untreated hypertension with :
* Clinical indication for an ABPM
* Clinical indication for a frailty measurement

Exclusion Criteria:

* Opposition to the use of data
* Inability to perform ABPM

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 75 years old, admitted for consultation or day hospitalisation in the Geriatric Service of the CHRU, living at home, with treated or untreated hypertension with clinical indication for an ABPM and Clinical indication for a frailty measurement
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Standard deviation of 24 hours Systolic Arterial blood pressure | From inclusion until 24 hours
  Assessed on 24-hour Arterial Blood Pressure Measurement (ABPM)

SECONDARY OUTCOMES:
Coefficient of variation of 24 hours systolic Arterial blood pressure | From inclusion until 24 hours
  Assessed on 24-hour Arterial Blood Pressure Measurement (ABPM)
Standard deviation of 24 hours Diastolic Arterial blood pressure | From inclusion until 24 hours
  Assessed on 24-hour Arterial Blood Pressure Measurement (ABPM)
Standard deviation of 24 hours Pulse arterial blood pressure | From inclusion until 24 hours
  Assessed on 24-hour Arterial Blood Pressure Measurement (ABPM)
Standard deviation of 24 hours Mean arterial blood pressure | From inclusion until 24 hours
  Assessed on 24-hour Arterial Blood Pressure Measurement (ABPM)
Coefficient of variation of 24 hours Diastolic Arterial blood pressure | From inclusion until 24 hours
  Assessed on 24-hour Arterial Blood Pressure Measurement (ABPM)
Coefficient of variation of 24 hours Pulse arterial blood pressure | From inclusion until 24 hours
  Assessed on 24-hour Arterial Blood Pressure Measurement (ABPM)
Coefficient of variation of 24 hours Mean arterial blood pressure | From inclusion until 24 hours
  Assessed on 24-hour Arterial Blood Pressure Measurement (ABPM)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD-PhD, Study Chair — CHRU de NANCY
Locations (1):
- CHRU de NANCY, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No